CLINICAL TRIAL: NCT01533441
Title: Study of the Effect of Food Vitamin K2 Intake in Association With a Fermented Dairy Product on Patients Treated With Vitamin K Antagonist (VKA)
Brief Title: Vitamin K2 Intervention in Patients With Vitamin K Antagonists
Acronym: SAFEK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Danisco (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: SAFE K study
Record Dates: First submitted 2012-02-03; First posted 2012-02-15 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Thrombosis
Keywords: anticoagulant therapy; INR; vitamin K2; vitamin K antagonist
MeSH Terms: conditions — Thrombosis | interventions — Vitamin K 2; Vitamin K 1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- placebo low VKA (Placebo Comparator)
  Interventions: Dietary Supplement: Vitamin K2
- Placebo high VKA (Placebo Comparator): Microcrystalline cellulose
  Interventions: Dietary Supplement: Vitamin K2
- Vitamin K2 Low VKA (Active Comparator)
  Interventions: Dietary Supplement: Vitamin K2
- Vitamin K2 high VKA (Active Comparator)
  Interventions: Dietary Supplement: Vitamin K2

INTERVENTIONS:
Dietary Supplement: Vitamin K2 — 4 months retrospective period and 4 months dairy product + treatment (vitaminK2 or placebo) intervention
  Other Names: phylloquinone,; menaquinone

SUMMARY:
The objective of the SAFE K study is to demonstrate that in patients treated with the antagonists of vitamin K (VKA), a daily intake of vitamin K2 (75 micrograms/day) as naturally produced by the ferments used in fermented dairy products, does not upset the balance of anticoagulant treatment.Fifty-two patients will be chosen to receive either verum or placebo for four months after a 4-month run-in period.In addition, the study evaluates if regular consumption of vitamin K2 reduce the need of changing the dose of anticoagulation treatment and improve the markers of bone mineralisation.

DETAILED DESCRIPTION:
Randomisation of the study subjects will be done by two randomisation lists depending on whether the dose of VKA is high or low. Randomisation will be balanced and stratified depending on the average dose of VKA before the inclusion in order that each arm would have the same number of patients receiving a dose lower than the used anticoagulant treatments.

The level of vitamin K intake will be determined during the study visits using dietary questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* treated with anticoagulants
* INR range between 2-3
* TTR (time in therapeutic range)equal or higher 56% during the 4 months before the inclusion

Exclusion Criteria:

* consumption of significant amounts of products conatining vitamin K
* regular consumption of dietary supplements susceptible to contain vitamin K
* milk intolerant or refusing a daily consumption of dairy product
* previous insufficient earlier therapeutic VKA follow-up
* cardiac, renal or severe respiratory insufficiency, diseases interfering fat absorption, significant abnormalities in safety parameters, clinically significant thrombotic or hemorrhagic event

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
INR | change from baseline at two months
  Prothrombin time
INR | change from baseline at four months
  prothrombin time

SECONDARY OUTCOMES:
c/uc osteocalcin ratio | change from baseline at two months
  immunoassay method
FVII from plasma | change from baseline at two months
  chronometric method
FII | change from baseline at two months
  chronometric method
Plasma vitamin K levels | change from base-line at two months
  HPLC
c/uc osteocalcin ratio | change from baseline at four months
  immunoassay method
FVII | change from baseline at four months
  chronometric method
FII | change from baseline at four months
  chronometric method
Plasma vitamin K level | change from baseline at four months
  HPLC

CONTACTS AND LOCATIONS:
Overall Officials: Kirsti Tiihonen, PhD, Study Director — Danisco Sweeteners Oy; Ludovic Drouet, Professor, Study Chair — IVS/CREATIF, Hopital Lariboisiere; Claire Bal dit Sollier, Study Chair — IVS/CREATIF, Hopital Lariboisiere
Locations (1):
- Unite de Recherches Therapeutiques, Hopital Lariboisiere, Paris, France